CLINICAL TRIAL: NCT00324376
Title: A Randomized, Cross-Over Study to Compare Once A Day Sevelamer Dosing With Three Times Per Day Sevelamer Dosing
Brief Title: Study to Compare Once A Day Sevelamer Dosing With Three Times Per Day Sevelamer Dosing
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GTC-68-209
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sevelamer

INTERVENTIONS:
Drug: Sevelamer hydrochloride

SUMMARY:
A randomized, cross-over, open-label study will be conducted to evaluate the equivalency, safety and tolerability of sevelamer once per day dosing, given with the largest meal, compared with standard three times per day dosing, in hemodialysis patients previously using sevelamer. Following a two week Run-In period, a total of 24 patients will be randomized to one of the following treatment sequences:

1. sevelamer dosed once a day with the largest meal followed by standard three times per day dosing with meals
2. sevelamer dosed three times per day with meals followed by once a day dosing with the largest meal. Patients will maintain a fixed daily dose throughout both treatment periods based on the most recently prescribed sevelamer dose prior to screening.

ELIGIBILITY:
Inclusion Criteria:

* life expectancy of at least 12 months,
* patients have received hemodialysis three times per week for 3 months or longer,
* patients maintained on sevelamer in a daily dose of ≤ 9,600 mg as their only phosphate binder with serum phosphorus concentrations at the last two measurements between 3.0 and 6.5 mg/dL (0.97 and 2.10 mmol/L).

Exclusion Criteria:

* active bowel obstruction,
* dysphagia,
* swallowing disorders,
* severe gastrointestinal motility disorders,
* active ethanol or drug abuse (excluding tobacco),
* need for antidysrhythmic or antiseizure medications used to control these conditions,
* poorly controlled diabetes mellitus or hypertension,
* active vasculitis,
* active malignancy other than basal-cell carcinoma,
* HIV infection,
* any clinically significant unstable medical condition as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2003-03; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Treatment compared on basis of serum phosphorus at end of each treatment and calcium corrected for albumin,calcium-phosphorus product,albumin,iPTH,total,LDL,HDL,non-HDL cholesterol,triglycerides. Safety evaluated on AEs;change in lab values.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (2):
- United States (2):
  - Renal Care Group, Olympia Fields, Illinois
  - Kidney and Hypertension Center, Cincinnati, Ohio

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Fishbane S, Delmez J, Suki WN, Hariachar SK, Heaton J, Chasan-Taber S, Plone MA, Moe S. A randomized, parallel, open-label study to compare once-daily sevelamer carbonate powder dosing with thrice-daily sevelamer hydrochloride tablet dosing in CKD patients on hemodialysis. Am J Kidney Dis. 2010 Feb;55(2):307-15. doi: 10.1053/j.ajkd.2009.10.051. Epub 2009 Dec 30. PMID 20042256